CLINICAL TRIAL: NCT02596412
Title: MINIDOCS : Contribution of Augmented Reality to Reduce Pain During of Botulinum Toxin Injections in Cerebral-palsied Children. A Randomized Controlled Trial
Brief Title: Augmented Reality to Reduce Pain During Botulinum Toxin Injections in Cerebral-palsied Children
Acronym: MINIDOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Fondation Apicil (Other); Fondation Motrice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL15-043-1
Record Dates: First submitted 2015-10-30; First posted 2015-11-04 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy
Keywords: children; botulinum toxin; augmented reality; Pain
MeSH Terms: conditions — Cerebral Palsy; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- augmented reality (Mini-Docs) on tablet (Experimental): • Cerebral-palsied children using the module with augmented reality (Mini-Docs) on tablet during TB injections in addition to regular drug techniques (experimental group)
  Interventions: Other: use the module with augmented reality (Mini-Docs) on tablet during TB injection
- Control (No Intervention): Cerebral-palsied children with the usual pain care during TB injections, which combines drug techniques to distractibility techniques (control group)

INTERVENTIONS:
Other: use the module with augmented reality (Mini-Docs) on tablet during TB injection — Provision of a tablet with a module using augmented reality (Mini-Docs) during TB injections in addition to the commonly used drug technology
  Arms: augmented reality (Mini-Docs) on tablet

SUMMARY:
Children with cerebral palsy may benefit from treatment with botulinum toxin injections to decrease spasticity for improve function and quality of life. These injections cause repeated pain throughout childhood and may be the cause of post-traumatic stress despite drug and non-drug pain management. The Mini-Docs project of the French Red Cross has a module based on a digital device with augmented reality. Distracting the child, the use of this module on a tablet would reduce pain felt during botulinum toxin injections.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of the use of a module with augmented reality (Mini-Docs) on pain during botulinum toxin injections in children with cerebral palsy aged from 3 to 8 years

Method: Randomized controlled trial comparing a group of children receiving the module with augmented reality of the Mini-Docs and drug pain management (nitrous oxide and medications), with a group of children receiving the usual care of pain management that combines drug pain management (nitrous oxide and medications) and distraction techniques. The device with the augmented reality module allows the child to add virtual content to the real images of the care. The pain will be assessed for each child 10 minutes after the injections, using a self-assessment scale (the Faces Pain Scale - Revised) or a heteroevaluation scale (the Face Legs Activity Cry Consolability scale given by the nurse). The study will be conducted in two centers of physical medicine and pediatric rehabilitation of the French Red Cross (Paris and Lyon).

Expected Results:

* Decreasing children's pain during botulinum toxin injections
* Decreasing anxiety in children and parents during injections
* Increasing coping skills in children
* Facilitating of the achievement of the therapeutic goal during injections

ELIGIBILITY:
Inclusion Criteria:

* Cerebral-palsied children, whose diagnosis of cerebral palsy was confirmed by a neurologist reported in the medical record
* Aged 3 to 8 years (until the day before 9 years old)
* With a functional level of Gross Motor Function Classification System (GMFCS) I, II, III or IV
* Treated by TB injection (child with or without a history of TB injections)
* With a sufficient level oral expression to respond to questionnaires and to interact with the nurse for the use of augmented reality device
* Obtaining written parental consent and oral approval by the child

Exclusion Criteria:

* Impossibility to assess pain during the session by the FLACC scale or FPS-R scale
* Visual disturbances excluding to use of the augmented reality device
* Severe cognitive impairment making it possible to answer questionnaires
* Child of functional level child GMFCS V
* Child with a specific request for distraction (eg if the child demands to watch a cartoon). This in order not to interfere with the coping strategies used by the child.
* Refusal on the part of the parents to sign consent, and refusal on the part of child to use the tablet
* Child not benefiting from social security coverage

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Pain during botulinum toxin (TB) injections | Assessment 10 minutes after TB injection
  Standardized pain scores will be calculated on a scale from 0 to 10 points using validated tools adapted to the age of the child: the Faces Pain Scale - Revised (FPS-R) and the Face Legs Activity Cry Consolability (FLACC). With each scale, patient scoring ≥ 4 is defined as painful.

SECONDARY OUTCOMES:
Level of anxiety of cerebral palsied children before TB injection | Assessment up to 1h before TB injection and up to 1h after TB injection
  measured by the Modified Yale Preoperative Anxiety Scale Questionnaire (m-Ypas), completed by the parents accompanying the child before and after TB injections
Level of parental anxiety accompanying the child during care | Assessment up to 1h before TB injection and up to 1h after TB injection
  It will be measured by the Stait Trait Anxiety Inventory (STAI) questionnaire before and after TB injections.
Assessment of Mini-Docs acceptability | 7 days after TB injection
  Mini-Docs acceptability will be assessed by telephone interview with the parents of the intervention group 7 days after the of TB injection

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie LUCET, Principal Investigator — Centre Médecine Physique et de Réadaptation pour Enfants de Bois-Larris - Croix-Rouge française
Locations (2):
- France (2):
  - Centre Médecine Physique et de Réadaptation pour Enfants de Bois-Larris - Croix-Rouge française, Lamorlaye
  - Centre Médico-Chirurgical de Réadaptation des Massues - Croix-Rouge française, Lyon